CLINICAL TRIAL: NCT01806233
Title: Lu' Acupuncture and Moxibustion Treatment on Ischemic Stroke
Brief Title: Lu's Acupuncture and Moxibustion Treatment on Stroke
Acronym: LAMTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3534123123
Record Dates: First submitted 2013-02-26; First posted 2013-03-07 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Ischemic Stroke; Paralysis
MeSH Terms: conditions — Ischemic Stroke; Paralysis | interventions — Acupuncture Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): acupuncture
  Interventions: Procedure: Acupuncture
- Rehabilitation (Experimental): rehabilitation exercise
  Interventions: Procedure: Rehabilitation

INTERVENTIONS:
Procedure: Acupuncture — The treatment group：60 patients receive Acupuncture ，selecting acupoint on:Shenting（DU24), Baihui（DU20）, Fengchi（GB20), Hanyan（GB4）, Jianyu（LI15）, Quchi（LI11）,Waiguan（SJ5）, Zusanli（ST36）, Fenglong（ST40）, Xingjian(LV2), Yongquan（KI1）, 20minutes each time，ten times / treatment course，two treatment courses in total.
  Arms: Acupuncture
Procedure: Rehabilitation — The matched group：60 patients receive rehabilitation treatment，45 minutes each once，ten time as a period of treatment，two periods of treatment in all.
  Other Names: Rehabilitation treatment
  Arms: Rehabilitation

SUMMARY:
There will be successive changes in traditional Chinese medicine rehabilitation for stroke patients with limb hemiparetic through therapy of acupuncture and moxibustion.

DETAILED DESCRIPTION:
There will be difference in stroke outcomes of ischemic stroke patients with limb hemiparetic from acute to chronic phase under Lu' acupuncture and moxibustion.

ELIGIBILITY:
Inclusion Criteria:

* The ages of stroke patients from 40 years old to 70 years old.
* The principle diagnosis according to <diagnosis-treatment criteria of stroke(trial implementation)>formulated by Collaboration Acute Brain Diseases of State Administration of Traditional Chinese Medicine in 1996；Ischemic stroke confirmed by CT brain or MRI brain,with stable medical condition and awareness clear.
* Recent stroke from 7 days to 6 months after onset.
* Stroke with limb movement disorder and hypomyotonia，NIHSS≤10，ASHWORTH≤1，GCS>8.
* Written informed consent by inpatient.

Exclusion Criteria:

* Stroke with conscious disturbance or serious cognitive impairment.
* Stroke with limb spasm；ASHWORTH≥1.
* Having cardiac pacemaker，metallic foreign body in treatment position，or hemorrhagic tendency.
* Being oversensitive to electrical stimulus.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-03; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Simplified Fugl-Meyer Scale | 8 weeks
  5 times a week, last 4 weeks,assessment on 4 weeks and 8 weeks

SECONDARY OUTCOMES:
Burden of Stroke Scale-Boss | 6 months
  5 times a week, last 4 weeks,assessment on 8 weeks and 6 months
Modified Barthel Index | 6 months
  5 times a week, last 4 weeks,assessment on 8 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, MD, Study Chair — Shanghai University of Traditional Chinese Medicine; Yi Wu, MD, Study Chair — Huashan Hospital; Jie Jia, MD, Study Director — Huashan Hospital; Yi Song, MM, Study Director — Shanghai University of Traditional Chinese Medicine; Zouqin Huang, MM, Principal Investigator — Shanghai University of Traditional Chinese Medicine; Xiaoxin You, MM, Principal Investigator — Shanghai University of Traditional Chinese Medicine; Qinhui FU, MD, Principal Investigator — Shanghai University of Traditional Chinese Medicine; Jun Wang, MM, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital,Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Pei J, Fu QH, Zhan YJ. The Prognostic Value of Traditional Chinese Medicine Symptoms in Acute Ischemic Stroke: A Pilot Study. Evid Based Complement Alternat Med. 2020 Jul 15;2020:1520851. doi: 10.1155/2020/1520851. eCollection 2020. PMID 32733577